

# NON-INTERVENTIONAL (NI) STUDY PROTOCOL

# **Study Information**

| Title | Comparative Effectiveness of Tumor<br>Necrosis Factor (TNF) inhibitors and<br>Tofacitinib, overall, by line of therapy and<br>by combination therapy |
|---|---|
| Protocol Number | A3921389 |
| Protocol Version Identifier | 2.0 |
| Date | 18 April 2022 |
| Active Substance | L04AA29 |
| Medicinal Product | Xeljanz (tofacitinib immediate release (IR) and extended release (XR)) |
| Research Question and Objectives | <ol> <li>The objectives of this study are as follows:</li> <li>To compare the effectiveness of tofacitinib and TNFs at 6 months and 12 months, overall and stratified by mono- and combination therapy.</li> <li>To investigate the association between line of tofacitinib therapy and response at 6 and 12 months.</li> </ol> |
| Author | PPD<br>PPD |

This document contains confidential information belonging to Pfizer. Except as otherwise agreed to in writing, by accepting or reviewing this document, you agree to hold this information in confidence and not copy or disclose it to others (except where required by applicable law) or use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Pfizer must be promptly notified.

# 1. TABLE OF CONTENTS

| 1. TABLE OF CONTENTS | 2 |
|---|---|
| 2. LIST OF ABBREVIATIONS | |
| PPD | |
| 4. ABSTRACT | 7 |
| 5. AMENDMENTS AND UPDATES | |
| 6. MILESTONES | 9 |
| 7. RATIONALE AND BACKGROUND | 9 |
| 8. RESEARCH QUESTION AND OBJECTIVES | 9 |
| 9. RESEARCH METHODS | 10 |
| 9.1. Study Design | 10 |
| 9.2. Setting. | 10 |
| 9.2.1. Inclusion Criteria | 10 |
| 9.2.2. Exclusion Criteria | 11 |
| 9.3. Variables | 11 |
| 9.4. Data Sources | 12 |
| 9.5. Study Size | 13 |
| 9.6. Data Management | 13 |
| 9.6.1. Record Retention | 13 |
| 9.7. Data Analysis | 14 |
| 9.8. Quality Control | 14 |
| 9.9. Limitations of the Research Methods | 15 |
| 9.10. Other Aspects | 15 |
| 10. PROTECTION OF HUMAN SUBJECTS | 15 |
| 10.1. Patient Information | 15 |
| 10.2. Patient Consent. | 15 |
| 10.3. Institutional Review Board (IRB)/Independent Ethics Committee (IEC) | 15 |
| 10.4. Ethical Conduct of the Study | 15 |
| 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS | 16 |
| 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS | |
| 13. REFERENCES | 17 |

| Xeljanz (tofacitinib) |
|--------------------------------------------|
| A3921389 NON-INTERVENTIONAL STUDY PROTOCOL |
| Protocol Amendment 1 18 April 2022 |

| 14. LIST OF TABLES | 18 |
|----------------------------------------|----|
| 15. LIST OF FIGURES | 18 |
| ANNEX 1. LIST OF STAND ALONE DOCUMENTS | 18 |
| ANNEX 2. ADDITIONAL INFORMATION | 18 |

# 2. LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|--------------|-------------------------------------------|
| ACR | American College of Rheumatology |
| AE | Adverse Event |
| BMI | Body Mass Index |
| CABG | Coronary Artery Bypass Grafting |
| CCP | Cyclic Citrullinated Peptide |
| CDAI | Clinical Disease Activity Index |
| CHF | Congestive Heart Failure |
| COPD | Chronic Obstructive Pulmonary Disease |
| CRP | C-reactive Protein |
| csDMARD | Conventional Synthetic Disease Modifying |
| | Antirheumatic Drug |
| CV | Cardiovascular |
| DAS | Disease Activity Score |
| DMARD | Disease Modifying Antirheumatic Drug |
| ESR | Erythrocyte Sedimentation Rate |
| EQ-5D | European Quality of Life-5 Dimensions |
| FDA | Food and Drug Administration |
| HAQ | Health Assessment Questionnaire |
| HEOR | Health Economics and Outcomes Research |
| ID | Identification |
| IEC | Independent ethics committee |
| IL | Interleukin |
| ILD | Interstitial Lung Disease |
| IR | Immediate Release |
| IRB | Institutional Review Board |
| JAK | Janus Kinase |
| mACR | Modified American College of Rheumatology |
| MD | Doctor of Medicine |
| mHAQ | Modified Health Assessment Questionnaire |
| MI | Myocardial Infarction |
| MOA | Mechanism of Action |
| MTX | Methotrexate |
| NI | Non-interventional |
| NSAID | Nonsteroidal Anti-inflammatory Drug |
| PASS | Post Authorization Safety Study |
| PCI | Percutaneous Coronary Intervention |
| RA | Rheumatoid Arthritis |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| TIA | Transient Ischemic Attack |

| Abbreviation | Definition |
|--------------|-----------------------|
| TNF | Tumor Necrosis Factor |
| US | United States |
| VAS | Visual Analogue Scale |
| XR | Extended Release |

Xeljanz (tofacitinib) A3921389 NON-INTERVENTIONAL STUDY PROTOCOL Protocol Amendment 1, 18 April 2022

# 4. ABSTRACT

Not applicable.

# **5. AMENDMENTS AND UPDATES**

| Amendment<br>number | Date | Protocol<br>section(s)<br>changed | Summary of amendment(s) | Reason |
|---|---|---|---|---|
| 1 administrative | 18 April<br>2022 | 6 Milestones | Milestones were updated. | The planned milestones were adjusted to align with information in sponsor's internal systems. |

#### 6. MILESTONES

| Milestone | Planned date |
|--------------------------|------------------|
| Start of data collection | 31 January 2021 |
| End of data collection | 30 November 2021 |
| Final study report | 30 October 2022 |

#### 7. RATIONALE AND BACKGROUND

Rheumatoid arthritis (RA) is a chronic and systemic inflammatory disease with an estimated prevalence of 0.5-1.0% and a mean annual incidence of 0.02-0.05% within Western populations. RA is characterized by inflammation, joint destruction, and progressive disability. Joint destruction is frequently irreversible resulting in significant cumulative morbidity. Patients experience a broad range of co-morbidities. These patients are also treated with multiple classes of agents, including nonsteroidal anti-inflammatory drugs (NSAIDs), glucocorticoids, and disease modifying antirheumatic drugs (csDMARDs) including biologicals, each of which carry significant risks as well as benefits.

Tofacitinib is the first oral janus kinase (JAK) inhibitor to show clinical efficacy in the management of RA. Many of the cytokines that are dysregulated in RA signal through JAKs.<sup>2,3,4</sup> Tofacitinib reduces the production of proinflammatory mediators<sup>5</sup> by inhibiting the signaling of multiple cytokines important in the pathogenesis of RA. Unlike biological therapies, such as tumor necrosis factor (TNF) inhibitors and anti-interleukin (IL)-6 receptor monoclonal antibodies that markedly inhibit one cytokine pathway over an extended period of time, JAK inhibition by tofacitinib results in a pattern of partial and reversible inhibition of the intracellular effects from several inflammatory cytokines.

This study will help demonstrate if there has been a shift in the treatment landscape between 2016 (time of the last Corrona registry analysis of this type) and 2020, in regards to tofacitinib use in earlier lines of therapy and use as monotherapy. We hope to gain a more current understanding of comparative effectiveness of the two mechanisms of action (MOA) in clinical practice.

#### 8. RESEARCH QUESTION AND OBJECTIVES

There are two primary objectives for this study:

- 1. To compare the effectiveness of tofacitinib and TNFs at 6 months and 12 months, overall and stratified by mono- and combination therapy.
- 2. To investigate the association between line of tofacitinib therapy and response at 6 and 12 months.

#### 9. RESEARCH METHODS

## 9.1. Study Design

To meet the study objectives, an observational retrospective cohort study will be conducted using patients enrolled in the Corrona RA Registry initiating to facitinib on or after November 2012. Patients receiving to facitinib or TNF after failing a csDMARD (2<sup>nd</sup>-4<sup>th</sup> line patients) will be included to assess the comparative effectiveness of to facitinib and TNF (stratified by monotherapy and combination therapy) as well as the impact of line of therapy on the effectiveness of to facitinib.

For further details, please refer to the detailed Statistical Analysis Plan (SAP) included as a stand alone document.

## 9.2. Setting

The Corrona RA Registry is a prospective, multicenter, observational disease-based registry launched in 2001. This registry contains clinical data (eg, disease activity scores, laboratory results, comorbidities, imaging results, patient-reported outcomes data, etc.) that is not available in claims databases. The current Corrona dataset includes 189 private and academic active clinical sites with over 817 providers throughout 42 states in the US. This registry collects data from both the providers and the patients at the time of a regular office visit. Corrona has enrolled over 54,000 patients with RA. The collection of data from Corrona represents over 195,750 patient years of data.

To be included in the Corrona RA Registry, patients must be at least 18 years of age and have a diagnosis of RA by a rheumatologist. Patients are excluded from the registry if they are unable or unwilling to provide informed consent. The inclusion/exclusion criteria for this particular analysis are described in Sections 9.2.1 and 9.2.2.

#### 9.2.1. Inclusion Criteria

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

- 1. RA patients in Corrona initiating tofacitinib <u>OR</u> a TNF biologic (adalimumab, etanercept, infliximab, golimumab, certolizumab pegol) after 06 November 2012 (market approval of Tofacitinib) during follow-up in Corrona with no prior use of tofacitinib. Only the patient's first initiation after 06 November 2012 will be included in the analysis.
- 2. Have a 6 and/or 12-month follow-up visit (with +/-2 month window).
- 3. Have Clinical Disease Activity Index (CDAI) measures at baseline and at the follow-up visit.

#### 9.2.2. Exclusion Criteria

Patients meeting any of the following criteria will not be included in the study:

1. Patients who have not failed methotrexate (MTX) or another csDMARD (ie, 1<sup>st</sup> line initiators).

#### 9.3. Variables

## Patient characteristics at baseline:

- Gender, age, race, and ethnicity.
- Duration of RA (Age at onset).
- Comorbidity history:
  - Cardiovascular disease: Myocardial Infarction (MI), stroke, Transient Ischemic Attack (TIA), acute coronary syndrome, coronary artery disease, congestive heart failure (CHF), revascularization procedure including percutaneous coronary intervention (PCI), coronary artery bypass grafting (CABG) or coronary artery stents, ventricular arrhythmia, cardiac arrest, unstable angina, other cardiovascular (CV) events, carotid artery disease;
  - Hypertension;
  - Chronic Obstructive Pulmonary Disease (COPD);
  - Asthma;
  - Interstitial Lung Disease (ILD)/Pulmonary Fibrosis;
  - Diabetes mellitus;
  - Serious infections;
  - Cancer: lung cancer, breast cancer, lymphoma, skin cancer (melanoma, basal, squamous), and other cancer;
  - Thromboembolic events: deep vein thrombosis, peripheral arterial thromboembolic and pulmonary embolism.
- C-reactive Protein (CRP).
- Erythrocyte Sedimentation Rate (ESR).
- Serum positive (Rheumatoid factor/Cyclic Citrullinated Peptide (CCP)).

- Smoking status.
- Work status.
- Height, weight, and body mass index (BMI).
- Insurance (patient reported).
- Prednisone use.

#### **Disease activity measures:**

- Physician reported:
  - CDAI:
  - MD global assessment;
  - Tender and swollen joint count (28);
  - Disease Activity Score (DAS) 28;
  - Modified American College of Rheumatology (mACR) 20/50/70.
- Patient reported:
  - Health Assessment Questionnaire (HAQ);
  - mHAQ;
  - Patient global assessment;
  - Patient pain VAS;
  - Patient fatigue VAS;
  - Morning stiffness.

### 9.4. Data Sources

Patients are enrolled in the Corrona RA Registry during regularly-scheduled office visits. Upon enrollment, providers complete a set of Enrollment Questionnaires, including a 28 joint count on RA patients. Patients also complete an Enrollment Questionnaire, which captures several data elements, including the Health Assessment Questionnaire (HAQ) and the European Quality of Life-5 Dimensions (EQ-5D). Both patient and provider reported disease activity measures obtained at each visit are captured in Corrona; this includes tender and swollen joint counts (28 joint counts), patient and physician global disease assessment,

patient pain assessment and HAQ scores. Providers and patients complete Follow-Up Questionnaires approximately every six months. During the course of a regularly-scheduled office visit, the provider performs assessments as mandated on the Corrona Provider Questionnaires with recording of pertinent data. Results from certain laboratory tests are included, but not mandated. Likewise, during regularly-scheduled office visits, patients are asked to complete Questionnaires designed to capture information ranging from their general demographics and experience with prescription drug use to an overall global assessment of their disease. Early Follow-Up visits occur and questionnaires are completed whenever a registry patient is being prescribed or receiving a first dose of a new (different) *eligible medication* at a routine office visit. Eligible medications are biologics, biosimilars, and JAK inhibitors Food and Drug Administration (FDA) approved for the treatment of RA. The next regularly scheduled visit is calculated from the previous visit. Data are collected on patients for as long as they consent to remain in the study.

## 9.5. Study Size

We used significance level of 0.05 (p=0.05), 80% power (80% rejecting the null hypothesis), and two independent sample equal-variance t-test for power calculation. The null hypothesis is no difference in mean of CDAI measure between treatment groups.

Previous study using Corrona RA registry data shown standard deviation (SD) is about 14 which will be used to estimate the sample size. Using software, it is estimated that 342 subjects would be needed in each of the treatment groups in order to detect a statistically significant difference in mean CDAI of 3 between the two groups. Increasing the mean of CDAI difference to 6, would require 87 patients in each group.

Current feasibility within the registry is 1,383 to facitinib patients (588 monotherapy patients and 795 combination patients) so the necessary sample size has been achieved.

#### 9.6. Data Management

All statistical analyses will be performed using STATA Version 15.1 (StataCorp, LLC, College Station, TX). All analyses will be carried out under the direction of Dr. Ying Shan of Corrona.

#### 9.6.1. Record Retention

To enable evaluations and/or inspections/audits from regulatory authorities or Pfizer, Corrona agrees to keep all study-related records, including safety reporting forms, source documents, detailed records of treatment disposition, and adequate documentation of relevant correspondence (eg, letters, meeting minutes, and telephone call reports). The records should be retained by Corrona according to local regulations or as specified in the vendor contract, whichever is longer. Corrona must ensure that the records continue to be stored securely for so long as they are retained.

If Corrona becomes unable for any reason to continue to retain study records for the required period, Pfizer should be prospectively notified. The study records must be transferred to a designee acceptable to Pfizer.

Study records must be kept for a minimum of 15 years after completion or discontinuation of the study, unless Corrona and Pfizer have expressly agreed to a different period of retention via a separate written agreement. Records must be retained for longer than 15 years if required by applicable local regulations.

Corrona must obtain Pfizer's written permission before disposing of any records, even if retention requirements have been met.

## 9.7. Data Analysis

Detailed methodology for summary and statistical analyses of data collected in this study will be documented in a statistical analysis plan (SAP), which will be dated, filed and maintained by the sponsor. The SAP may modify the plans outlined in the protocol; any major modifications of primary endpoint definitions or their analyses would be reflected in a protocol amendment.

## 9.8. Quality Control

Corrona or its designee monitors the conduct of the registry at each investigative site. Monitoring is primarily conducted remotely. Onsite monitoring visits are conducted once every three years, as needed, or as requested. A review of registry records including, but not limited to, the informed consent forms, Questionnaires, original source documents such as supporting medical records and office notes, subject study files, and any other registry documentation is conducted in accordance with applicable regulatory guidelines and the protocol. Corrona and its designees are required to maintain the confidentiality of all subjects during and after an on-site monitoring visit.

Quality control checks are built into the on-screen data entry systems in an attempt to reduce queries and provide immediate feedback to the investigator regarding inadvertent omissions and out of range or noncompliant values. Changes made at any time are recorded in an audit trail that includes the date, time, and electronic identification (ID) of the person making the change.

Corrona will address and resolve discrepancies by requesting clarifications and/or missing data from the investigator as needed. Each investigator is expected to designate a point of contact to address such inquiries and to promptly address and resolve issues. Representatives or designees from Corrona reserve the right to perform random or systematic audits of Corrona Questionnaires at an investigator's site in order to assess the accuracy of the reported data compared to the information contained in the original medical records.

#### 9.9. Limitations of the Research Methods

The Corrona RA Registry includes a sample of adults with RA that are not necessarily representative of all adults with RA in the US. In particular, these are RA patients with clinical visits with rheumatologists. Patients are recruited by rheumatologists who are required to indicate diagnosis upon enrollment of the patient into the Corrona RA Registry. In addition, history of medication use prior to enrollment is derived from what is reported by patients and their current rheumatologist within the registry. Since registry reporting is not based on a fixed visit schedule, exact timing of visits to fit 6, 12, 24, or 36 months of post index data is not available for all patients so windows of time are used to determine eligible visits. The "cause" of visits is not captured, although the assumption can likely be made that the rheumatologist visit is "RA related." The registry captures provider reported prescribing; there are no measures of patient adherence.

As this is real world study, missing data could be expected for demographic characteristics (eg, age, etc.); however, the number of patients with missing data is expected to be very small. With multiple time points, some visits may have missing CDAI

## 9.10. Other Aspects

Not applicable.

#### 10. PROTECTION OF HUMAN SUBJECTS

#### 10.1. Patient Information

This study involves data that exist in anonymized structured format and contain no patient personal information.

#### 10.2. Patient Consent

As this study involves anonymized structured data, which according to applicable legal requirements do not contain data subject to privacy laws, obtaining informed consent from patients by Pfizer is not required.

## 10.3. Institutional Review Board (IRB)/Independent Ethics Committee (IEC)

There must be prospective approval of the study protocol, protocol amendments, and other relevant documents (eg, informed consent forms if applicable) from the relevant IRBs/IECs. All correspondence with the IRB/IEC must be retained. Copies of IRB/IEC approvals must be forwarded to Pfizer.

## 10.4. Ethical Conduct of the Study

The study will be conducted in accordance with legal and regulatory requirements, as well as with scientific purpose, value and rigor and follow generally accepted research practices described in Good Practices for Outcomes Research issued by the International Society for Pharmacoeconomics and Outcomes Research (ISPOR).

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

This study involves data that exist as structured data by the time of study start. In these data sources, individual patient data are not retrieved or validated, and it is not possible to link (ie, identify a potential association between) a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (AE) (ie, identifiable patient, identifiable reporter, a suspect product, and event) cannot be met.

#### 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

For all publications relating to the Study, Pfizer will comply with recognized ethical standards concerning publications and authorship, including Section II - "Ethical Considerations in the Conduct and Reporting of Research" of the Uniform Requirements for Manuscripts Submitted to Biomedical Journals, http://www.icmje.org/index.html#authorship, established by the International Committee of Medical Journal Editors.

In the event of any prohibition or restriction imposed (eg, clinical hold) by an applicable competent authority in any area of the world, or if party responsible for collecting data from the participant is aware of any new information which might influence the evaluation of the benefits and risks of a Pfizer product, Pfizer should be informed immediately.

#### 13. REFERENCES

- 1. Alamanos Y, Drosos AA. Epidemiology of adult rheumatoid arthritis. Autoimmun Rev 2005;4(3):130-6.
- 2. Walker JG, and Smith MD. The Jak-STAT pathway in rheumatoid arthritis. J Rheumatol, 2005;32(9):1650-3.
- 3. McInnes IB, Schett G. Cytokines in the pathogenesis of rheumatoid arthritis. Nat Rev Immunol 2007; 7(6):429-42.
- 4. McInnes IB, Schett G. The pathogenesis of rheumatoid arthritis. N Engl J Med 2011; 365(23):2205-19.
- 5. Meyer DM, Jesson MI, Li XO, et al. Anti-inflammatory activity and neutrophil reductions mediated by the JAK1/JAK3 inhibitor, CP-690,550, in rat adjuvant-induced arthritis. J Inflamm 2010; 7:41.

# 14. LIST OF TABLES

None.

# **15. LIST OF FIGURES**

None.

# ANNEX 1. LIST OF STAND ALONE DOCUMENTS

| Number | Date | Title |
|---|---|---|
| 1 | 09 September<br>2020 | Comparative Effectiveness of TNFs and tofacitinib, overall and by combination therapy |
| 2 | 09 September 2020 | Comparative Effectiveness of Tofacitinib by Line of Therapy |

# **ANNEX 2. ADDITIONAL INFORMATION**

Not Applicable.

# **Document Approval Record**

| Document Name: | A3921389 Non Interventional Study Protocol Amendment 1 (clean) 18<br>Apr2022 |
|---|---|
| Document Title: | A3921389 Non Interventional Study Protocol Amendment 1 (clean) 18<br>Apr2022 |

| Signed By: | Date(GMT) | Signing Capacity |
|------------|----------------------|------------------|
| PPD | 21-Apr-2022 18:45:17 | Final Approval |